CLINICAL TRIAL: NCT06926101
Title: MARGINAL BONE LEVELS AROUND IMPLANTS PLACED BY PARTIAL OR FULL-THICKNESS FLAP: A 3-YEAR RANDOMIZED CONTROLLED CLINICAL TRIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Antonino Palazzolo, DDS, MSc, MClindDent (Oral Surgery), PhD, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1564/19
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Dental Implant; Dental Implant Therapy; Edentulism
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implant placement through partial thickness flap procedure (Experimental)
  Interventions: Device: dental implants
- Implant placement through full thickness flap procedure (Active Comparator)
  Interventions: Device: dental implants

INTERVENTIONS:
Device: dental implants — dental implant placement by full or partial thickness flap

SUMMARY:
Each enrolled patient received one implant placed with the partial-thickness flap disconnect mode (PT Test Group) or the full-thickness flap disconnect mode (FT Control Group) from the same implant system (Anyridge, MegaGen Implant Co., Gyeongbuk, South Korea). Each implant was placed at 0.5 mm sub-crest as per protocol guidelines. This choice was made according to the current scientific literature. This implant system has specific macrostructural and microstructural techniques that allow high levels of standards. The fixture-abutment connection is internally conical at 2.8 mm with 5° indexing: this feature makes it possible to reduce the prosthetic microgap, move the platform away from the bone margin while maintaining an optimal crestal margin and prevent rotation or unscrewing of the prosthetic component. Each implant was placed at 1 mm sub-crest as per protocol guidelines. This choice was made according to the current scientific literature.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years of age; 2. Need for implant placement therapy in the posterior area (from the second premolar to the second molar) due to a failing tooth; 3. Presence of adjacent and opposing natural teeth; 4. Sufficient mesial-distal and interocclusal space for placement of the implant and definitive restoration; 5. Sufficient apical bone to achieve a minimum primary stability of 30Ncm.

Exclusion Criteria:

* 1. Diagnosis of periodontal disease; 2. Medical or general contraindications for the surgical procedure, such as systemic diseases, history of head and neck radiation therapy, current steroid treatment, neurological or psychiatric conditions affecting oral hygiene, immune-compromised status, severe clenching, or bruxism; 3. Heavy smoking (>10 cigarettes/day); 4. Active infection at the implant site.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
marginal bone levels | each year up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinic University of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No